CLINICAL TRIAL: NCT05447065
Title: Impact of Vitamin D Supplementation on COVID-19 Vaccine Response and IgG Antibodies in Deficient Women.
Acronym: CoVıD-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Avrasya University (Other)
Responsible Party: Principal Investigator, Fatih Cesur, Assistant Professor, Avrasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021/02; 2021/02 (Other Grant/Funding Number: Avrasya University)
Record Dates: First submitted 2022-07-05; First posted 2022-07-07 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: COVID-19 Pandemic; D Vitamin Deficiency; Antibody Hypersensitivity
Keywords: COVID-19 Vaccine; Antibody; IgG; D vitamin; Nutrition
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants using vitamin D supplements (Experimental): Participants in the experimental group were given 150,000 IU (10 ml) of vitamin D3 supplementation, and it was used regularly for 2 months. From the first measurement, 2 more measurements were taken, 28 days apart, and a total of 3 measurements were taken from the participants.
  Interventions: Dietary Supplement: Vitamin D supplement
- Participants not using vitamin D supplements (No Intervention): No supplement was given to the control group. From the first measurement, 2 more measurements were taken, 28 days apart, and a total of 3 measurements were taken from the participants.

INTERVENTIONS:
Dietary Supplement: Vitamin D supplement — Only the experimental group (D) received the vitamin D supplement.
  Arms: Participants using vitamin D supplements

SUMMARY:
Decreased immunity in individuals causes a decrease in vaccine response, and vitamin D worsens this course. Vitamin D is thought to be a vitamin that can strengthen the innate immune response, inhibit the adaptive system, and modulate the vaccine response.

The effect of vitamin D intake on antibodies was studied.

ELIGIBILITY:
Inclusion Criteria:

* The study consisted of young volunteer women who completed 2 doses of COVID-19 vaccines, did not receive the 3rd dose, and spent an average of 65 days over the 2nd dose. Participants were included in the study when IgM value was negative, IgG value was positive, they were not older than 25 years, and serum 25-Hydroxy (25(OH)) vitamin D was below 30 ng/mL.

Exclusion Criteria:

* In addition, individuals participating in the research who were pregnant, had physician-diagnosed cardiovascular diseases, had kidney or liver failure, and had the chronic obstructive pulmonary disease were not included in the study.

Ages: 19 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-05-07 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
From the first measurement, 2 more measurements were taken, 28 days apart, and a total of 3 blood measurements were taken from the participants. Antibody levels were measured with the fluorescent immunological (FIA) method. | Within research completion, an average of 8 week
  Compared to other coronaviruses, it was understood that there is an instant need for a vaccine to prevent SARS CoV-2 because of its faster transmission. However, it is very important to determine that the COVID-19 vaccine is immune to individuals, and it has been emphasized that Immunoglobulin G (IgG) levels are checked for immune testing and it is important that these levels are high. People's immune systems or nutritional levels are influential in the high rate or efficiency of immunoglobin levels Studies have reported that individuals with adequate and balanced nutrition have a stronger immune system

SECONDARY OUTCOMES:
From the first measurement, 2 more measurements were taken, 28 days apart, and a total of 3 blood measurements were taken from the participants. 25(OH) Vitamin D level levels were measured with the fluorescent immunological (FIA) method. | Within research completion, an average of 8 week
  Since a treatment process is not clear at the beginning of the COVID-19 disease, these supplements, such as vitamin D, C, and B vitamin groups and zinc minerals, have been given to COVID-19 patients in the clinic. In addition, 25-Hydroxy(25(OH)) vitamin D deficiency is a common condition for these patients. Accordingly, skeletal system diseases, immune system diseases, inflammatory bowel diseases, respiratory tract infections, viral infections, etc. affect situations are also seen. The pathogenesis relationship of 25(OH) vitamin D with the COVID-19 pandemic is consistently seen in the clinical data. In addition, 25(OH) vitamin D deficiency has a negative effect on people with COVID-19. For this reason, it is thought that hospitalizations due to COVİD-19 are increasing In a way, it is claimed to be an important factor in the severe course of the disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Avrasya University, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Derived] Cesur F, Atasever Z, Ozoran Y. Impact of vitamin D3 supplementation on COVID-19 vaccine response and immunoglobulin G antibodies in deficient women: A randomized controlled trial. Vaccine. 2023 Apr 24;41(17):2860-2867. doi: 10.1016/j.vaccine.2023.03.046. Epub 2023 Mar 27. PMID 37003908
- See also: Related Info — https://doi.org/10.3389/fimmu.2019.00065
- See also: Related Info — https://doi.org/10.1016/J.RETRAM.2022.103344
- See also: Related Info — https://doi.org/10.1093/AJCN/77.1.204
- See also: Related Info — https://doi.org/10.1016/j.jsbmb.2021.105964

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-06-05): https://cdn.clinicaltrials.gov/large-docs/65/NCT05447065/SAP_000.pdf